CLINICAL TRIAL: NCT04685148
Title: Short Time Oestrogen as a Candidate Strategy to Prevent Postpartum Depression in a High-risk Group: a Randomised, Placebo-controlled Trial.
Brief Title: Maternal Mental Health Trial
Acronym: MAMA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vibe G Frøkjær, MD, PhD (Other)
Collaborators: Herlev Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor-Investigator, Vibe G Frøkjær, MD, PhD, Sponsor-investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-001592-33
Record Dates: First submitted 2020-12-16; First posted 2020-12-28 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder; Postpartum Depression
Keywords: Postpartum period; Mother-infant interaction; Personalised prevention; Perinatal depression; Hormone sensitivity; Estradiol
MeSH Terms: conditions — Depressive Disorder, Major; Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Estradiol patches (200 μg per day) 0-3 weeks postpartum.
  Interventions: Drug: Transdermal patch estradiol
- Placebo (Placebo Comparator): Placebo patches (Coloplast Comfeel) for 0-3 weeks postpartum
  Interventions: Drug: Transdermal patch placebo

INTERVENTIONS:
Drug: Transdermal patch estradiol — Estradiol patches (200 μg per day by transdermal delivery) will be administered at day 0 (+1) to day 21 postpartum.
  Arms: Intervention
Drug: Transdermal patch placebo — Placebo patches will be administered at day 0 (+1) to day 21 postpartum.
  Arms: Placebo

SUMMARY:
Perinatal depression affects 10-15% of women postpartum and has a recurrence rate of 40%. Women who develop perinatal depression might be particularly susceptible to the rapid and large changes in sex steroid hormones, particularly estradiol, across pregnancy to postpartum. This trial aims 1) to evaluate the preventive effect of transdermal estradiol treatment in the immediate postpartum on depressive episodes in a subgroup of women at high-risk for perinatal depression, and 2) to determine if a set of biomarker gene transcripts can identify this subgroup and thus form the basis for future personalised prevention or treatment.

The MAMA Trial is a double-blind, 1:1 randomised, placebo-controlled trial. The trial involves maternity wards at three university hospitals in the Capital Region of Denmark. Women who are singleton pregnant in the third trimester with a prior history of perinatal depression are eligible to participate. Participants will be randomised to either estradiol patches (200 μg per day) or placebo patches for three weeks starting immediately postpartum.

The primary statistical analysis will be performed based on the intention-to-treat principle. A sample size of 220 will provide the trial with 80% power (alpha 0.05, beta 0.2) to detect a reduction in postpartum depression of 50% and to tolerate a drop-out of around 20%.

DETAILED DESCRIPTION:
Major depressive disorder affects twice as many women as men. Women are at increased risk for depression in life phases, where endogenous sex steroid hormone milieu changes; such as in puberty, during late pregnancy to postpartum and across menopausal transition. This includes a subtype of MDD, perinatal depression (PND) that affects 10-15% of mothers postpartum and has a recurrence rate of 40% in subsequent pregnancies. PND is a disabling disorder that affects the entire family, including development and future health of the infant.

The underlying risk and resilience mechanisms in MDD are far from clear, consequently, current treatment strategies are suboptimal. Women who develop PND might be particularly sensitive to the rapid and large changes in sex steroid hormone milieu, seen in the transition from high levels of sex steroid hormones, in particular estradiol, in pregnancy to low levels in the hormone withdrawal phase postpartum. Thus, PND is most likely has a distinct pathophysiology, which may provide a unique opportunity for protecting mental health by targeted short-term prevention in the immediate postpartum period.

Intriguingly, recent human data has provided direct evidence for sex hormone manipulation to provoke subclinical depressive symptoms in about 12% of healthy volunteers. The phenomenon was linked to changes in estradiol, which were induced by the pharmacological manipulation with a Gonadotrophin Releasing Hormone agonist. Estradiol affects critical domains and key brain regions known to be dysfunctional in women with major depressive disorder. Estradiol sensitivity predisposes to PND, which can be demonstrated at the level of gene transcription in clinical cohorts, and is also directly supported by recent research results. Such peripheral markers of estradiol sensitivity may prove useful in identifying individuals at excess risk for PND, also in their first pregnancy, and thus may help direct preventive efforts for the women who can benefit the most.

Transdermal estradiol emerges as a promising preventive treatment option for the postpartum onset of PND supported by epidemiological, preclinical, and clinical research, robust and rapid response to estradiol in some pilot postpartum depression (PPD) trials with few side effects and minimal breastmilk passage to the infant. Further, transdermal estradiol appears to be effective in preventing clinically significant depressive symptoms among perimenopausal women, which is another group of women in hormonal transition phase.

Previously, a double-blind randomized, controlled trial (RCT) showed effect of treatment with transdermal estradiol on manifest PND. A recent pilot RCT with transdermal estradiol as a candidate treatment for postpartum depression failed to achieve its primary outcome, but notably, did reduce depressive symptoms postpartum compared to placebo.

Rather than treating manifest depressive episodes postpartum, the investigators here propose a different approach: to target, and potentially prevent, early risk mechanisms in the first three weeks postpartum, and to direct this preventive strategy towards women in high risk. This immediate and early postpartum timing corresponds to the peak risk period and covers the peak of hormonal decline postpartum.

This trial aims 1) to evaluate the preventive effect of transdermal estradiol treatment in the immediate postpartum on depressive episodes in a subgroup of women at high risk for Perinatal Depression with postpartum onset, and 2) to determine if a set of biomarker gene transcripts can identify this subgroup and thus form the basis for future personalized prevention or treatment.

Methods The Maternal Mental Health (MAMA) Trial is designed as a double-blind, 1:1 randomized, placebo-controlled superiority trial setting involving maternity wards at three university hospitals in the Capital Region of Denmark.

Women who are singleton pregnant in third trimester with a prior history of perinatal depression (onset before six months postpartum) and aged 18 to 45 years are eligible to participate.

The women will be assessed for eligibility by the midwife or obstetrician when attending antenatal care at the outpatient clinic. Eligible participants who verbally consent to receive more information about the trial will subsequently be contacted by telephone. Written informed consent is obtained before inclusion in the MAMA Trial.

The randomisation will be conducted by the capital region pharmacy. Trial participants, clinical care providers, research assistants, investigators, outcome assessors, and data analysists will all be blinded to allocation.

The investigators calculated that a sample of 2*88 complete cases would provide the trial with 80% power (at a two-sided alpha level of 0.05) to detect a reduction in postpartum depression of 50%. Thus, with a study number of 2*110, the design is considered solid and can tolerate 22% dropouts.

The primary statistical analysis will be performed on basis of the intention-to-treat principle. The investigators will compare data on the primary outcome for the two groups for the superiority of estradiol over placebo with Pearson's chi-squared test.

Secondary outcomes with a continuous distribution will be compared between groups with respect to the mean (Student's t-test) if the distribution is unimodal and symmetric, or to the median if the distribution is unimodal but asymmetric, or otherwise to the ranks of the observations (Mann-Whitney test). A test on the difference in proportions will be used for binary secondary outcomes and a Pearson's chi-squared test will be used for categorical data.

As a sensitivity analysis, we will use an instrumental variable approach to estimate causal treatment effect using randomisation as an instrument.

Ethical considerations The short-term administration of estradiol transdermally is not expected to pose unacceptable or intolerable side-effects, disrupt breastfeeding or pass to the infant in any dosages that may pose a risk to the infant. Should un-expected side effects for mother or infant occur or be suspected, the treatment will be disrupted immediately. When removing the patch, serum concentrations of estradiol return to baseline levels within 24 hours. Participants who develop levels of mental distress or depressive symptoms that approach clinical thresholds will be referred to relevant and timely psychiatric care by a trained clinician. All potentially sensitive personal data will be anonymized. The trial will adhere closely to the Helsinki declaration.

Prospect There is a pressing need to develop a preventive strategy to depressive episodes during pregnancy and childbirth, that is targeted, cheap, short-term, and easy to implement. Such work holds promise to positively affect women's mental health, their families, and importantly, if successful, may also improve long-term outcomes of the infant's physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnant
* Prior history of perinatal depression
* Age between 18 and 45 years

Exclusion Criteria:

* Moderate to severe depression with onset during pregnancy
* Severe psychiatric disorders (e.g. disorders with psychotic symptoms, schizophrenia, bipolar disorders, inpatient eating disorders and inpatient obsessive-compulsive disorders)
* Previous suicide attempts without having a depressive episode
* Prior history or ongoing neurological disorders (e.g. migraine or epilepsy)
* Severe somatic illness
* Prior history or ongoing cancer
* Prior history of venous thromboembolism, myocardial infarction, cerebrovascular thromboembolism or thrombophilia, or other risk factors clinically assessed after thrombophilia screening
* Deep vein thrombosis or pulmonary embolism in current pregnancy
* Pregnancy-induced hypertension or preeclampsia
* Pre-existing atherosclerosis or well-known cardiovascular risk factors (e.g. diabetes, hypertension)
* Other contraindication for oestrogen treatment (e.g. acute liver failure, severe varicose veins)
* Use of psychotropic pharmacology, except for short-term sleep support treatment
* Non-fluent in Danish or pronounced vision or hearing loss
* Body Mass Index (BMI) >35 kg/m2
* Ongoing alcohol or drug abuse
* Severe postpartum haemorrhage (>1500 ml)
* Severe illness in the infant or perinatal death

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Major Depression Disorder | 0-6 months postpartum
  Clinical diagnosis assessed by DSM-V criteria

SECONDARY OUTCOMES:
EPDS Depressive symptoms | 8-10 weeks postpartum
  Edinburgh Postnatal Depression Scale score. Score range: 0-30.
HamD6 Depressive symptoms | 8-10 weeks postpartum
  Score on the Hamilton 6-item depression scale. Score range 0-22.
Maternal mental wellbeing | 8-10 weeks postpartum
  WHO-5 Well-Being Index. Score range 0-100. Low score means less well-being.
Maternal anxiety | 8-10 weeks postpartum
  State Trait Anxiety inventory (STAI) score. Score range 20-80.
Parental stress | 8-10 weeks postpartum
  Parental Stress Scale. Score range 18-90.
Parental reflective capacity | 8-10 weeks postpartum
  Parental Reflective Functioning Questionnaire. Score range 12-60.
Parental competences | 8-10 weeks postpartum
  Parenting Sense of Competence scale. Score range 16-96.
Proportion of women who exclusively breastfeed their infants | 8-10 weeks postpartum
  Questionnaire developed for the trial. Categorical outcome.
Predictive value of composite gene transcription and DNA methylation marker for estrogen sensitivity | 8-10 weeks postpartum
  116 a priori defined gene transcripts, which where differentially expressed in third trimester of women who later developed perinatal depression with postpartum onset relative to pregnant women who did not and to other depressed (reference Mehta et al, 2014, Psychological Medicine, Mehta et al. 2018 British Journal of Psychiatry).
Maternal sleep quality | 8-10 weeks postpartum
  Pittsburgh Sleep Quality Index. Score range 0-21.
Maternal attachment to unborn child | Baseline time point at third trimester, i.e. week 34-37 of pregnancy
  Maternal Antenatal Attachment Scale. Score range 19-95.
Cold cognitive function | 8-10 weeks postpartum
  A later variable derived from simple reaction time test, Rey's Auditory Verbal Learning Task (Declarative memory, RAVLT), Letter-Number Sequence (Working Memory, LNS), and Intra-Extra Dimensional Set Shifting (Cognitive flexibility, IED, error rate)
Hot cognitive function | 8-10 weeks postpartum
  A latent variable derived from emotional Intensity Morphing Test (EIMT) and Infant Emotion Test (Maternal Distress Sensitivity and Infant Emotion Detection (IET)
Socio-emotional infant development | 8-10 weeks
  Ages and Stages questionnaire Social-emotional 2 (ASQ:SE-2) total score. Score range 0-160. Higher scores worse outcome.
Infant development (Bayley-III) | 8-10 weeks postpartum
  Cognitive, language and motor development score from Bayley-III test
Cortisol dynamics Cortisol dynamics | 3-5 weeks postpartum
  Cortisol awakening response in saliva (area under the curve with respect to increase from 0 to 60 minutes from awakening)
Cortisol evening Cortisol dynamics | 3-5 weeks postpartum
  Cortisol concentration in evening saliva from home sampling
Hair cortisol level Cortisol dynamics | 0-1 days postpartum
  Provides an estimate of cortisol exposure up to 6 months prior to delivery
Epigenetic markers relevant for infant HPA axis | 0-1 days postpartum
  FKBP5 methylation index
Estradiol level | 3 weeks postpartum
  Estradiol level in peripheral blood
Change in estradiol level | From baseline (third trimester of pregnancy) to 3 weeks postpartum
  Estradiol change pre- to postpartum in peripheral blood
Progesterone level | 3 weeks postpartum
  Progesterone level in peripheral blood
Change in progesterone level | From baseline (third trimester of pregnancy) to 3 weeks postpartum
  Progesterone change pre- to postpartum in peripheral blood
Allopregnanolone level | Baseline time point at third trimester, i.e. week 34-37 of pregnancy
  Allopregnanolone level in peripheral blood
Allopregnanolone level | 3 weeks postpartum
  Allopregnanolone level in peripheral blood
Change in allopregnanolone level | From baseline (third trimester of pregnancy) to 3 weeks postpartum
  Allopregnanolone change pre- to postpartum in peripheral blood
Negative bias in responses to infant vocalisations and video | 8-10 weeks
  Composite measure of negative bias score of ratings of 50 infant vocalisations and negative emotional expression.
Estradiol level | Baseline time point at third trimester, i.e. week 34-37 of pregnancy
  Estradiol level in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Vibe Gedsø Frøkjær, MD, PhD, Principal Investigator — Neurobiology Research Unit, copenhagen University hospital, Rigshospitalet, Denmark
Locations (1):
- Neurobiology Researc hUnit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
When the planned analyses from the trial are published, the data will become publicly available. According to the Danish legislation, data will be available only by approval by the Danish Data Protection Agency and with a signed agreement.
Supporting Information: Study Protocol
Time Frame: We expected that data will come available December 2026 and be available for approx. 4 years.
Access Criteria: Data will be available on reasonable request with approval by the Danish Data Protection Agency and with a signed agreement.

REFERENCES:
- [Derived] Hogh S, Hegaard HK, Renault KM, Cvetanovska E, Kjaerbye-Thygesen A, Juul A, Borgsted C, Bjertrup AJ, Miskowiak KW, Vaever MS, Stenbaek DS, Dam VH, Binder E, Ozenne B, Mehta D, Frokjaer VG. Short-term oestrogen as a strategy to prevent postpartum depression in high-risk women: protocol for the double-blind, randomised, placebo-controlled MAMA clinical trial. BMJ Open. 2021 Dec 30;11(12):e052922. doi: 10.1136/bmjopen-2021-052922. PMID 35763351